CLINICAL TRIAL: NCT01305707
Title: Continuation Electroconvulsive Therapy Associated With Pharmacotherapy Versus Pharmacotherapy Alone for Relapse Prevention in Major Depression. A Clinical, Controlled, Prospective and Randomized Trial
Brief Title: Continuation Electroconvulsive Therapy (C-ECT) for Relapse Prevention in Major Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties in recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Mikel Urretavizcaya Sarachaga, Psychiatrist, MD, PhD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TECHUB2007
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Depression
Keywords: Consolidation ECT; Pharmacotherapy; Efficacy; Depression; Prevention; Electroconvulsive therapy; Drug therapy
MeSH Terms: conditions — Depression | interventions — Drug Therapy; Antidepressive Agents; Venlafaxine Hydrochloride; Duloxetine Hydrochloride; Imipramine; Clomipramine; Nortriptyline; Sertraline; Fluoxetine; Citalopram; Paroxetine; Escitalopram; Mirtazapine; Mianserin; Antipsychotic Agents; Quetiapine Fumarate; Aripiprazole; Lithium; Clorazepate Dipotassium; Lorazepam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- C-ECT and Pharmacotherapy (Experimental): Consolidation treatment with ECT will be considered finished after 9 months of being started, at which time patients will stay only on the pharmacological treatment they already had. The study will be completed within 15 months of patient inclusion (six months after the end of C-ECT). Patient assessment and follow-up will be conducted by participant researchers. Blind rater will conduct clinical and adverse effects ratings. A neuropsychologist will conduct neuropsychological assessments.
  Interventions: Device: C-ECT
- Pharmacotherapy (Active Comparator): Pharmacotherapy will remain unchanged since the acute episode to the end of the study. Psychotropics will be obtained as usually from the National Health System and will be prescribed according to data sheet.
  Interventions: Drug: PHARMACOTHERAPY

INTERVENTIONS:
Device: C-ECT — C-ECT will be administered through a Thrymatron System IV device (Somatics, LLC, ISO 13485:2003). Electrode placement will be bilateral and energy administered during consolidation treatment will be same used in the acute episode. C-ECT will be given weekly for the first month, fortnightly for the following two months and monthly during the next 6 months. A total of 14 C-ECT sessions will be given over 9 months of treatment.
  Pharmacotherapy will remain unchanged since the acute episode to the end of the study. Drugs will be obtained as usually from the National Health System and will be prescribed according to data sheet and it will have a duration of 15 months.
  Other Names: Thrymatron System IV device (Somatics, LLC, ISO 13485:2003).; Pharmacotherapy:; Antidepressants:; - Venlafaxine 75-225 mg/d. N06AX16; - Duloxetine 60-120 mg/d. N06AX21; - Imipramine 100-300 mg/d. N06AA02; - Clomipramine 75-225 mg/d. N06AA04; - Nortriptyline 75-200 mg/d. 906AA10; - Sertraline 50-200 mg/d. N06AB06; -Fluoxetine 20-40 mg/d. N06AB03; - Citalopram 20-60 mg/d. N06AB04; - Paroxetine 20-40 mg/d. N06AB05; - Escitalopram 10-20 mg/d. N06AB10; - Mirtazapine 15-45 mg/d. N06AX11; - Mianserin 10-60 mg/d. 906AX03; - Trazadone 50-200 mg/d. 906AX05; - Reboxetin 2-12 mg/d. N06AX18; Antipsychotic drugs; - Olanzapine 2'5-20 mg/d. N05AH03; - Risperidone 0'5-9 mg/d. N05AX08; - Quetiapine 50-600 mg/d. N05AH04; - Aripiprazole 5-30 mg/d. N05AX12; Lithium: 200-1200 mg/d. 905AN01; Anxyiolitics:; - Diazepam 2'5-50 mg/d. N05BA01; - Clorazepate 5-50 mg/d. N05BA05; - Lorazepam 1-10 mg/d. N05BA06
  Arms: C-ECT and Pharmacotherapy
Drug: PHARMACOTHERAPY — Pharmacotherapy will remain unchanged since the acute episode to the end of the study. Psychotropics will be obtained as usually from the National Health System and will be prescribed according to data sheet and will have a 15 month duration.
  Other Names: Pharmacotherapy:; Antidepressants:; - Venlafaxine 75-225 mg/d. N06AX16; - Duloxetine 60-120 mg/d. N06AX21; - Imipramine 100-300 mg/d. N06AA02; - Clomipramine 75-225 mg/d. N06AA04; - Nortriptyline 75-200 mg/d. 906AA10; - Sertraline 50-200 mg/d. N06AB06; -Fluoxetine 20-40 mg/d. N06AB03; - Citalopram 20-60 mg/d. N06AB04; - Paroxetine 20-40 mg/d. N06AB05; - Escitalopram 10-20 mg/d. N06AB10; - Mirtazapine 15-45 mg/d. N06AX11; - Mianserin 10-60 mg/d. 906AX03; - Trazadone 50-200 mg/d. 906AX05; - Reboxetin 2-12 mg/d. N06AX18; Antipsychotic drugs; - Olanzapine 2'5-20 mg/d. N05AH03; - Risperidone 0'5-9 mg/d. N05AX08; - Quetiapine 50-600 mg/d. N05AH04; - Aripiprazole 5-30 mg/d. N05AX12; Lithium: 200-1200 mg/d. 905AN01; Anxyiolitics:; - Diazepam 2'5-50 mg/d. N05BA01; - Clorazepate 5-50 mg/d. N05BA05; - Lorazepam 1-10 mg/d. N05BA06
  Arms: Pharmacotherapy

SUMMARY:
OBJECTIVES:

To evaluate the comparative efficacy and security of Continuation Electroconvulsive Therapy associated with pharmacotherapy versus pharmacotherapy alone in the prevention of depressive relapse.

METHODS:

Demographic and clinical variables will be collected and side effects scales and neurocognitive battery will be performed. Variables of efficacy: relapse percentage in both groups in one year (primary variable); time without relapse. Main variable of security: occurrence of side effects and neurocognitive performance.

DESIGN: Randomized controlled clinical trial.

SAMPLE:

104 outpatients diagnosed with unipolar depression (DSM-IV-R criteria) who had remitted with a course of bilateral ECT. They will be randomized to two groups of treatment.

SETTING: Psychiatry Department at Bellvitge University Hospital.

ANALYSIS: Descriptive analysis of clinical variables; survive analysis and Cox model of regression.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a severe psychiatric disorder that affects more than 6 million people in our country and has a life prevalence of 8.9% for men and 16. 5% for women (Haro et al, 2007). Besides, in recent decades, its incidence is increasing (Kessler et al, 2004). MDD has high recurrence rates and 25% of the cases develop chronification. Moreover it can occur at any age leading to severe disability. The majority of studies published in this field demonstrated the efficacy of antidepressant treatment in a short or medium-term basis, but there is a lack of long-term clinical trials regarding antidepressant efficacy and published ones present methodological problems. At present, a line of fundamental research in therapeutics includes pragmatic studies because they can answer crucial and specific questions in clinical practice. Therefore, the aim of this project is to conduct a pragmatic, parallel, randomized trial with 2 treatment arms to answer a key question of great interest to psychiatrists: Is it more effective to extend the use of ECT as maintenance therapy (together with drug therapy) rather than just using drug therapy in patients that previously required an acute ECT course for a depressive episode? This study is a controlled randomized clinical trial that starts after the remission of the acute depressive episode. Once patients have clinically remitted they will be randomized in two groups:

1. C-ECT together with pharmacotherapy (same treatment used in the acute episode).
2. Maintenance pharmacotherapy treatment (same treatment used in the acute episode).

Consolidation treatment with ECT will be considered finished after 9 months of being started, at which time patients will stay only on the pharmacological treatment they already had. The study will be completed within 15 months of patient inclusion (six months after the end of C-ECT). Patient assessment and follow-up will be conducted by participant researchers. Blind rater will conduct clinical and adverse effects ratings. A neuropsychologist will conduct neuropsychological assessments.

ELIGIBILITY:
Inclusion Criteria:

* MDD diagnosis by DSM IV-TR.
* ECT requirement during acute episode. Therapeutic indication will be based on clinical criteria, following APA guidelines. During the acute episode, patients will be controlled by the usual clinical care team.
* Complete clinical remission (HDRS < or = 7 across two weeks).
* Appropriate intellectual level that allows adequate communication.
* Women of childbearing potential must use contraceptive methods.
* Signed Consent form.
* Other axis I or II diagnosis by DSM-IV-TR, except for nicotine dependence.
* To be in maintenance ECT program.
* To receive ECT during the previous three months of the acute episode.
* Pregnancy or breastfeeding.

Exclusion Criteria:

* Other axis I or II diagnosis by DSM-IV-TR, except for nicotine dependence.
* To be in maintenance ECT program.
* To receive ECT during the previous three months of the acute episode.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale 21 items (HDRS-21) | One year. HDRS will be assessed in each follow-up visit (weekly the first month, fortnightly the second and third month, monthly the following 6 months and quarterly at 12 and 15 months).
  HDRS-21 will measure the relapse year in each group. Relapse will be defined as the reappearance of relevant symptoms after resolutin of the acute episode, measured by a scoring in HDRS-21 between 15-17 over two following measures or a HDRS>18 score in a single measure.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE 35) | Basal, at 8 months and 12 months
  Assessment of general cognitive status.
UKU - Adverse effects rating scales | Every assessment (weekly, fortnightly, monthly and quarterly) till the month 15 of the follow-up.
  Qualitiative measure of side effects in each treatment group.
Demographical Data Memory (MEDABI-20) | Basal, at 8 months and 12 months
  Descriptive measure of cogntive status.
Rey Figure | Basal, at 8 months and 12 months
  Measure of visual perception, concentration and memory.
Trail Making Test A | Basal, at 8 months and 12 months
  Measure of attention and cognitive flexibility.
Trail Making Test B | Basal, at 8 months and 12 months
  Measure of attention and cognitive flexibility.
Stroop Test | Basal, at 8 months and 12 months
  Measure of selective attention, cognitive flexibility and processing speed as well as executive function.
Direct and inverse digits (WAIS, Weschler Adults Intelligence Sacle). | Basal
  Measure of general intelligence and attention
Vocabulary WAIS (Weschler Adults Intelligence Scale) | Basal
  Measure of general intelligence
Frequency Hospitalization Quotient | One year
  Measure of number of hospitalization per year.
Hospital Day Quotient (HDQ) | One year
  Number of days hospitalized per year.

CONTACTS AND LOCATIONS:
Overall Officials: Mikel Urretavizcaya Sarachaga, MD, PhD, Principal Investigator — Hospital Universitari de Bellvitge - IDIBELL; Èrika Martínez Amorós, MD, Principal Investigator — Corporacion Parc Tauli
Locations (3):
- Spain (3):
  - Hospital Universitari de Bellvitge, IDIBELL, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Corporació Sanitària Parc Tauli, Sabadell, Barcelona